CLINICAL TRIAL: NCT00138385
Title: A Randomized Comparison of the Immune Response to Either Inactivated or Live, Attenuated Influenza Vaccine in Children 5-9 Years of Age
Brief Title: Comparison of Inactivated and Live, Attenuated Influenza Vaccine in Children 5-9 Years of Age-Year 3 Amendment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04-079
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2007-11

CONDITIONS: Influenza
Keywords: inactivated, attenuated, influenza vaccine, FluMist, Fluzone
MeSH Terms: conditions — Influenza, Human | interventions — FluMist; Influenza Vaccines

INTERVENTIONS:
Biological: FluMist
Biological: Fluzone

SUMMARY:
The purpose of this study is to evaluate how young children's bodies learn to fight against flu infection and to see how vaccines may help to fight against the flu. This is a Phase 4, single-center, randomized study of the immune responses of 40 children, ages 5-9, given one of two licensed influenza vaccines (either inactivated vaccine given in an arm muscle or live, attenuated vaccine inhaled through the nose). Study procedures will include up to 3 blood samples. Participants will complete a diary to document any side effects experienced following the vaccination. Participants will return to the clinic for a visit on Day 7-9 and again 4-6 weeks following vaccination. Participants that have not been previously vaccinated will receive a 2nd dose of vaccine. A follow up telephone call will occur 8-10 weeks following vaccination. Total study participation will be up to 75 days.

DETAILED DESCRIPTION:
This is a Phase 4, single-center, randomized clinical trial of the immune responses of children given one of two licensed influenza vaccines (either inactivated vaccine given IM or live, attenuated vaccine given intranasally). This study will enroll 40 healthy children 5-9 years of age. Subjects will be randomized to receive either FluMist or Fluzone. FluMist is approved for children older than 5 years and Fluzone is also approved for a broader age indication starting at 6 months of age. Subjects who receive FluMist will have the vaccine administered intranasally by large particle aerosol, 0.25 mL per nostril. Subjects receiving Fluzone will receive 0.5 mL given intramuscularly into the non-dominant deltoid muscle. Children who have not previously been immunized against influenza will receive a second dose of vaccine 4 weeks after the first dose. Children who receive two doses of vaccine will remain on the study for 8-10 weeks. The primary objective of this study is to compare the effector B cell responses at Day7-9 and the CD4 and CD8 T-cell responses, memory B-cell and the serology responses at Day 28 post-immunization following administration of one of two different influenza vaccines. Researchers will evaluate any increases in the immune response (CD4, CD8, B cell and serology responses) Day 0 to Day 7-9 for T-cells and ASCs, and from Day 0-28 for memory B-cell and serology responses. NK-cell and homing studies will also be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 5-9 years of age.
* Parents willing to sign informed consent.
* Availability for follow-up for the planned duration of the study at least 4 weeks after last immunization.
* Acceptable medical history by screening evaluation and brief clinical assessment.

Exclusion Criteria:

* History of immunodeficiency.
* Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease; diabetes mellitus; moderate to severe kidney impairment.
* Household contact with immunodeficiency due to disease, medication or radiation.
* Child receiving aspirin therapy or aspirin-containing therapy.
* History of Guillain-Barré syndrome.
* Malignancy, other than squamous cell or basal cell skin cancer.
* Autoimmune disease.
* History of asthma or reactive airways disease.
* Chronic cardiovascular and pulmonary disorder.
* Chronic metabolic diseases (including diabetes), renal dysfunction or hemoglobinopathies requiring regular medical follow-up or hospitalization during the preceding year.
* Use of immunosuppressive medication. Corticosteroid nasal sprays are permissible.
* Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol.
* Inactivated vaccine 14 days prior to vaccination.
* Live, attenuated vaccines within 60 days of study.
* Use of investigational agents within 30 days prior to study.
* Receipt of blood products or immunoglobulin in the past 6 months.
* Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment.
* Acute febrile illness on the day of vaccination.
* Known allergies to any component of the vaccine, including thimerosal.
* History of allergy to eggs or egg products.
* Any condition that, in the opinion of the investigator, might interfere with study objectives.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40
Dates: Start 2005-08; Study Completion 2007-06

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States